CLINICAL TRIAL: NCT03003351
Title: Assessment of the Natural History and Treatment Outcomes for Patients With Fistula - a Pro- and Retrospective Cohort Study
Brief Title: Zurich Fistula Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Benjamin Misselwitz, Principal Investigator, University of Zurich
Other Study IDs: KEK-ZH-Nr. 2016-00367
Record Dates: First submitted 2016-12-19; First posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Fistula;Rectal; Fistula; Rectouterine; Fistula; Rectovesical; Fistulas Recto Vaginal; Crohn Disease
Keywords: Fistula; Cohort Study
MeSH Terms: conditions — Rectal Fistula; Fistula; Rectovaginal Fistula; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (2):
- Fistula: Patients with Fistulaê that are not caused by Crohn's disease
- Fistula and Crohn's disease: Patients with Fistulae that are caused by underlying Crohn's disease

SUMMARY:
This is a pro- and retrospective cohort study to evaluate the natural history and outcome of various treatment options of patients with fistula. At each clinical visit parameters describing activity of a fistula, potential underlying Crohn's disease, investigations as well as the current treatment will be entered into a database. Selected patients can also be contacted by phone in the form of a structured interview. Data will be analyzed to determine treatment outcomes, characterize the natural history as well as risk factors for complications of treatment and an unfavorable disease course. The same data will be obtained and analyzed retrospectively from patients who visited the clinic prior to January 2017.

DETAILED DESCRIPTION:
Fistulizing disease remains a frequent and severe problem for patients with Crohn's disease (CD). Life-time prevalence of fistula for patients with CD has been estimated to be 17 - 50% [1-5] with a cumulative incidence of 33% and 50% after 10 years and 20 years disease duration, respectively. These numbers have been confirmed by population-based studies [6, 7].

Patients with CD and fistula have a decreased quality of life. Reasons include perianal pain, discharge from the vagina, abdominal wall, perianal region and urinary tract infections. Fistula are frequently associated with abscess formation [8]. Unfortunately, surgical and medical treatment options for fistula for CD patients remain limited. Treatment with the tumor-necrosis factor (TNF) antibody infliximab remains the best medical treatment option available: At least temporary fistula closure is observed for 55% of treated fistula (compared to 12% for placebo). However, treatment success is frequently limited to a short time period of 3 month [9, 10]: 34% of all fistula patients experience recurrent fistula despite therapy [6] and successful treatment is limited to one third patients. For these reasons, up to 82% of all fistula need surgical treatment. Surgical options include non-cutting setons, application of fibrin glue as a "fistula plug", ligation of the intersphincteric fistula tract (LIFT) and reparative surgery including mucosal advancement flaps. However, surgical therapy for fistula patients can be complicated by slow wound healing, recurrent disease and additional problems [11].

Combined medical and surgical treatment for patients with fistula and CD can significantly improve clinical outcomes [12-15]. However, the best combination of clinical and surgical methods has yet to be determined [16]. Open questions include timing of seton removal and outcomes of the various surgical procedures for different patient groups.

At the University Hospital Zurich (USZ) the investigators recently started a combined surgical and gastroenterological clinic for patients with fistula. In the new clinic patients are seen by gastroenterologists and surgeons and the investigators are aiming for joint treatment decisions. Due to this combination of expertise and improved access to gastroenterological and surgical resources the investigators are expecting better treatment results for the patients and improved satisfaction for patients and referring physicians.

With the current study the investigators want to achieve the following objectives:

* Continuous monitoring of the quality of medical and surgical treatment
* Determining the outcome of various fistula therapies and calculating risk factors for a favorable and unfavorable outcome
* Understanding the natural history of perianal fistula and calculate risk factors for a favorable and unfavorable outcome.

The investigators are therefore proposing a pro- and retrospective database containing data regarding the clinical history, patient symptoms, examinations, lab values as well as other parameters. The database will be used for quality management regarding the daily work at USZ and to improve understanding regarding treatment options and the natural history of fistula. The investigators expect significant benefits for future patients from their analysis.

ELIGIBILITY:
Inclusion Criteria:

* Fistula
* written informed consent

Exclusion Criteria:

* age under 18
* retrospective analysis: documented rejection of clinical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with fistulae
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change in Perianal disease activity index (PDAI) | 6 months after intervention

SECONDARY OUTCOMES:
Change in Fistula Drainage assessment | 3, 6 & 12months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hellers G, Bergstrand O, Ewerth S, Holmstrom B. Occurrence and outcome after primary treatment of anal fistulae in Crohn's disease. Gut. 1980 Jun;21(6):525-7. doi: 10.1136/gut.21.6.525. PMID 7429313
- [Background] Michelassi F, Stella M, Balestracci T, Giuliante F, Marogna P, Block GE. Incidence, diagnosis, and treatment of enteric and colorectal fistulae in patients with Crohn's disease. Ann Surg. 1993 Nov;218(5):660-6. doi: 10.1097/00000658-199321850-00012. PMID 8239781
- [Background] Solomon MJ. Fistulae and abscesses in symptomatic perianal Crohn's disease. Int J Colorectal Dis. 1996;11(5):222-6. doi: 10.1007/s003840050051. PMID 8951512
- [Background] Allan A, Keighley MR. Management of perianal Crohn's disease. World J Surg. 1988 Apr;12(2):198-202. doi: 10.1007/BF01658054. No abstract available. PMID 3293326
- [Background] Bell SJ, Williams AB, Wiesel P, Wilkinson K, Cohen RC, Kamm MA. The clinical course of fistulating Crohn's disease. Aliment Pharmacol Ther. 2003 May 1;17(9):1145-51. doi: 10.1046/j.1365-2036.2003.01561.x. PMID 12752351
- [Background] Loftus EV Jr, Schoenfeld P, Sandborn WJ. The epidemiology and natural history of Crohn's disease in population-based patient cohorts from North America: a systematic review. Aliment Pharmacol Ther. 2002 Jan;16(1):51-60. doi: 10.1046/j.1365-2036.2002.01140.x. PMID 11856078
- [Background] Loftus EV Jr, Silverstein MD, Sandborn WJ, Tremaine WJ, Harmsen WS, Zinsmeister AR. Crohn's disease in Olmsted County, Minnesota, 1940-1993: incidence, prevalence, and survival. Gastroenterology. 1998 Jun;114(6):1161-8. doi: 10.1016/s0016-5085(98)70421-4. PMID 9609752
- [Background] Givel JC, Hawker P, Allan R, Keighley MR, Alexander-Williams J. Entero-enteric fistula complicating Crohn's disease. J Clin Gastroenterol. 1983 Aug;5(4):321-3. doi: 10.1097/00004836-198308000-00007. PMID 6886354
- [Background] Bell SJ, Kamm MA. Review article: the clinical role of anti-TNFalpha antibody treatment in Crohn's disease. Aliment Pharmacol Ther. 2000 May;14(5):501-14. doi: 10.1046/j.1365-2036.2000.00777.x. PMID 10792111
- [Background] Present DH, Rutgeerts P, Targan S, Hanauer SB, Mayer L, van Hogezand RA, Podolsky DK, Sands BE, Braakman T, DeWoody KL, Schaible TF, van Deventer SJ. Infliximab for the treatment of fistulas in patients with Crohn's disease. N Engl J Med. 1999 May 6;340(18):1398-405. doi: 10.1056/NEJM199905063401804. PMID 10228190
- [Background] Schwartz DA, Loftus EV Jr, Tremaine WJ, Panaccione R, Harmsen WS, Zinsmeister AR, Sandborn WJ. The natural history of fistulizing Crohn's disease in Olmsted County, Minnesota. Gastroenterology. 2002 Apr;122(4):875-80. doi: 10.1053/gast.2002.32362. PMID 11910338
- [Background] Hyder SA, Travis SP, Jewell DP, McC Mortensen NJ, George BD. Fistulating anal Crohn's disease: results of combined surgical and infliximab treatment. Dis Colon Rectum. 2006 Dec;49(12):1837-41. doi: 10.1007/s10350-006-0656-5. PMID 17041753
- [Background] Gaertner WB, Decanini A, Mellgren A, Lowry AC, Goldberg SM, Madoff RD, Spencer MP. Does infliximab infusion impact results of operative treatment for Crohn's perianal fistulas? Dis Colon Rectum. 2007 Nov;50(11):1754-60. doi: 10.1007/s10350-007-9077-3. Epub 2007 Sep 27. PMID 17899271
- [Background] Topstad DR, Panaccione R, Heine JA, Johnson DR, MacLean AR, Buie WD. Combined seton placement, infliximab infusion, and maintenance immunosuppressives improve healing rate in fistulizing anorectal Crohn's disease: a single center experience. Dis Colon Rectum. 2003 May;46(5):577-83. doi: 10.1007/s10350-004-6611-4. PMID 12792431
- [Background] Regueiro M, Mardini H. Treatment of perianal fistulizing Crohn's disease with infliximab alone or as an adjunct to exam under anesthesia with seton placement. Inflamm Bowel Dis. 2003 Mar;9(2):98-103. doi: 10.1097/00054725-200303000-00003. PMID 12769443
- [Background] Marzo M, Felice C, Pugliese D, Andrisani G, Mocci G, Armuzzi A, Guidi L. Management of perianal fistulas in Crohn's disease: an up-to-date review. World J Gastroenterol. 2015 Feb 7;21(5):1394-403. doi: 10.3748/wjg.v21.i5.1394. PMID 25663759
- [Background] Irvine EJ. Usual therapy improves perianal Crohn's disease as measured by a new disease activity index. McMaster IBD Study Group. J Clin Gastroenterol. 1995 Jan;20(1):27-32. PMID 7884173
- [Background] Sostegni R, Daperno M, Scaglione N, Lavagna A, Rocca R, Pera A. Review article: Crohn's disease: monitoring disease activity. Aliment Pharmacol Ther. 2003 Jun;17 Suppl 2:11-7. doi: 10.1046/j.1365-2036.17.s2.17.x. PMID 12786607
- [Background] Vaizey CJ, Carapeti E, Cahill JA, Kamm MA. Prospective comparison of faecal incontinence grading systems. Gut. 1999 Jan;44(1):77-80. doi: 10.1136/gut.44.1.77. PMID 9862829
- [Background] Harvey RF, Bradshaw JM. A simple index of Crohn's-disease activity. Lancet. 1980 Mar 8;1(8167):514. doi: 10.1016/s0140-6736(80)92767-1. No abstract available. PMID 6102236